CLINICAL TRIAL: NCT01327729
Title: Clinical Trial of the Efficacy, Dosing, Safety and Tolerability of Y- Shaped Pegylated Interferon (YPEG-IFNα-2a) Plus Ribavirin in Egyptian Patients With Untreated Chronic Hepatitis C
Brief Title: Y- Shaped Pegylated Interferon (YPEG-IFNα-2a) Plus Ribavirin in Egyptian Patients With Untreated Chronic Hepatitis C
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioGeneric Pharma (Industry)
Collaborators: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: prof. dr. mohamed karim, cairo university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHT00234
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Self Efficacy; Hepatitis C
Keywords: pegylated interferon; interferon; HCV; genotype 4
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- YPEG-IFN α-2a one week (Active Comparator): this arm will be treated with: YPEG-IFN α-2a 180mcg/ week for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks
  Interventions: Drug: pegylated interferon alpha 2a YPEG-IFN α-2a 180mcg
- YPEG-IFN α-2a Ten days (Active Comparator): this arm will be treated with: YPEG-IFN α-2a 180mcg/10 days for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks
  Interventions: Drug: pegylated interferon alpha 2a YPEG-IFN α-2a 180mcg
- YPEG-IFN α-2a two weeks (Active Comparator): The third group will be treated with:
  YPEG-IFN α-2a 180mcg/ 2 weeks for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks.
  Interventions: Drug: pegylated interferon alpha 2a YPEG-IFN α-2a 180mcg

INTERVENTIONS:
Drug: pegylated interferon alpha 2a YPEG-IFN α-2a 180mcg — YPEG-IFN α-2a 180mcg dose form: subcutaneous dosage : 180 mcg frequency every week or ten days or 2 weeks according to the group
  Other Names: YPEG-IFN α-2a 180mcg; YPEG; pegylated interferon

SUMMARY:
The objective is to assess the efficacy, dosing, safety and tolerance of Y- shaped pegylated interferon (YPEG-IFNα-2a) plus ribavirin in Egyptian patients with chronic hepatitis C and with no prior treatment for hepatitis C virus (HCV).

Methods: Randomized, Open-label trial, in 3 parallel groups (each of 100 patients)

DETAILED DESCRIPTION:
Methods: Randomized, Open-label trial, in parallel groups (each of 100 patients). Treatment will be given for 48 weeks (positive HCV by polymerase chain reaction (PCR) patients at 24 weeks will be considered non responders) and follow-up for 24 weeks. Total treatment and follow-up duration: 72 weeks. Enrollment duration: 18 months. Total trial duration: 2 years and 9 month, including trial analysis (carried out in the 6 months following the follow-up completion of the last patient). Total number of patients: 300. Precision around the expected efficacy rate (45% in intention-to-treat analysis) will be 9.6% (α = 0.05).

Primary objective: to assess the efficacy, dosing, safety and tolerability of Y- shaped pegylated interferon (YPEG-IFNα-2a) plus ribavirin in Egyptian patients with chronic hepatitis C and with no prior treatment for HCV.

Secondary objective: To assess the plasma level of the YPEG-IFNα-2a in the first 30 patients in each group, to ensure therapeutic plasma level of the drug at 2 hours, 6 hours, 10 hours, 24 hours, 3 days, 5 days, 7 days, 10 days, 14 days and 28 days.

Treatment strategy:

Three groups in which each group will include 100 patients.

The first group will be treated with:

YPEG-IFN α-2a 180mcg/week for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks.

The second group will be treated with:

YPEG-IFN α-2a 180mcg/10 days for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks.

The third group will be treated with:

YPEG-IFN α-2a 180mcg/ 2 weeks for 48 weeks. Ribavirin 15 mg/kg/day for 48 weeks. HCV RNA by PCR will be done at 24 weeks and negative PCR patients will continue treatment for another 24 weeks and PCR positive patients will be considered non responders and will be followed up.

Evaluation of the dose efficacy and side effects will be obtained at 4 weeks and 12 weeks of treatment, and any serious side effects or significant dose difference in early virological response in a group will lead to shift of this group to the dose 180 mcg/week.

Main outcome:

Viral clearance by qualitative HCV RNA based on PCR 24 weeks after the end of treatment.

Secondary outcomes:

Evaluation of HCV RNA at 12 and 24 weeks; changes in HCV RNA load during treatment; normalization of ALT during treatment and 24 weeks after the end of treatment; study of side effects; histological changes 24 weeks after the end of treatment: decrease by at least 1 point of the Metavir score.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 65 years
* Chronic hepatitis C defined as: HCV antibodies using a third generation test; HCV-RNA positive by PCR; liver biopsy in the past 12 months; METAVIR score of A1 and F0 or higher
* ALT > 1 ULN in the 24 weeks prior to inclusion (W-26; W-2)
* Patients never treated with ribavirin, Interferon or PEG-Interferon
* Normal albumin, prothrombin time > 60%; normal bilirubin
* Alpha-foeto-protein < 3 times the normal range for the laboratory reference
* HBs antigen negative
* Anti Bilharzial antibodies if positive rectal snip shall be done. The examination may be repeated after praziquantel treatment for those with a positive test
* Hemoglobin > 11g/dl, leucocytes > 3000/mm3, neutrophils > 1500/mm3, platelets > 100 000/mm3, blood creatinin < 1.4 mg/dl
* Normal TSH (subjects needing treatment to maintain TSH within a normal range may be included if other eligibility criteria are respected)
* Anti-nuclear antibodies < 1/160
* Fasting blood sugar between 70-115mg/dl ; if glucose intolerance or diabetes, HbA1C < 8.5%
* Normal ophthalmologic examination in patients with history of blood pressure and/or diabetes
* Effective contraception (IUD, diaphragm and spermicide, condoms and spermicides, oral contraceptive, progesterone implants (Norplant), medroxyprogesterone acetate (Depo-provera), tubal ligation, vasectomy) during the treatment period for females. No breastfeeding during the study period
* Signed informed consent

Exclusion criteria

* Other liver diseases associated with chronic hepatitis C: co-infection with hepatitis B (positive HBs antigen); hemochromatosis; alpha-1 anti-trypsin deficiency; Wilson disease; alcoholism-related liver disease; Gilbert disease
* Alcohol intake > 50g/day for males and 40 g/day for females
* Ongoing intravenous drug use
* Aggravated liver cirrhosis: history or presence of ascitis, oesophageal varicosis, liver encephalopathy
* Hepatocellular carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
viral clearance at 72 weeks | 72 weeks
  assessment of the efficacy, dosing, safety and tolerability of Y- shaped pegylated interferon (YPEG-IFNα-2a) plus ribavirin in Egyptian patients with chronic hepatitis C and with no prior treatment for HCV.

SECONDARY OUTCOMES:
interferon level | 12 weeks
  assessment of the plasma level of the YPEG-IFNα-2a in the first 30 patients in each group, to ensure therapeutic plasma level of the drug at 2 hours, 6 hours, 10 hours, 24 hours, 3 days, 5 days, 7 days, 10 days, 14 days and 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD, Principal Investigator — cairo university - Kasr alaini school of medicine; Mohamed Karim F Ashour, MD, Study Director — Cairo university- Kasr Alaini school of medicine
Locations (1):
- Kasr Alaini school of medicne, Cairo, Cairo Governorate, Egypt